CLINICAL TRIAL: NCT00013611
Title: A Phase III Multicenter Randomized Study of the Biological and Clinical Efficacy of Subcutaneous Recombinant, Human Interleukin-2 in HIV-Infected Patients With Low CD4+ Counts Under Active Antiretroviral Therapy (SILCAAT Amendment 4)
Brief Title: Interleukin-2 Plus Antiretroviral Therapy for HIV-Infected Patients With Low CD4+ Counts (SILCAAT Study)
Acronym: SILCAAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: DAIDS, NIAID
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0303M44961; 01-I-0126 (Other: NIAID); NCT00002421 (obsolete NCT alias)
Record Dates: First submitted 2001-03-24; First posted 2001-03-26 (Estimated); Results first posted 2010-12-13 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infection
Keywords: HIV; Proleukin; IL-2; Adult; HAART; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiretroviral therapy alone (No Intervention)
- Proleukin plus antiretroviral therapy (Experimental)
  Interventions: Drug: Proleukin

INTERVENTIONS:
Drug: Proleukin — Recombinant IL-2 was given at a dose of 4.5 MIU twice daily subcutaneously for 5 consecutive days every 8 weeks, in addition to antiretroviral therapy, for 6 cycles. After the first 6 cycles, additional cycles were given to either achieve or maintain the patient's CD4+ cell count goal.
  Other Names: recombinanat interleukin-2; rIL-2
  Arms: Proleukin plus antiretroviral therapy

SUMMARY:
This study will examine whether interleukin-2 (IL-2) plus antiretroviral therapy (ART) slows HIV disease progression in patients with low CD4+ T cell counts compared with patients taking ART alone. CD4+ T cells are a subset of lymphocytes-white blood cells that are part of the body's immune system. IL-2 is a protein that is naturally produced by lymphocytes. Given in intermittent cycles, IL-2 can raise CD4+ T cell counts in some HIV-infected patients taking antiretroviral drugs. This study will examine whether the increase in CD4+ T cells lowers the risk of AIDS-related illnesses and death.

HIV-infected patients 18 years of age and older with a viral load under 10,000 copies per milliliter and a CD4+ T cell count between 50 and 299 cells per cubic millimeter who are taking antiretroviral therapy and who have not previously received IL-2 therapy may be eligible for this study. Candidates will be screened with a medical history, physical examination, and blood and urine tests. Participation in the study will be from 4.5 to 6 years, depending on what point in the duration of the study the individual patient is enrolled.

Patients will be randomly assigned to receive IL-2 plus ART or ART alone. All participants will be advised individually about the best ART regimen for them. Patients in the IL-2 treatment group will be taught how to self-inject IL-2 under the skin (similar to insulin injections). They will inject IL-2 twice a day for 5 days every 8 weeks for the first year (until week 49 of the study). From week 49 on they may receive 5-day cycles of IL-2 every 4 months when needed to maintain CD4+ T cell count elevations. An extra cycle may be given 2 months after the week 49 follow-up visit (see follow-up schedule below), depending on their CD4+ T cell count. Patients whose cell counts have not increased after 12 to 16 months of IL-2 treatment will discuss with the doctor the possibility of stopping IL-2. Those who do stop IL-2 treatment will be asked to remain in the study for follow-up evaluations.

All patients will be followed in the clinic every 2 months for the first year of the study (weeks 1, 9, 17, 25, 33, 41 and 49) and every 4 months during years 2-6 for a brief history and physical exam, urine and blood tests, return of diary cards (record of drug side effects) and medication review. During the visits from the second year on, patients will also be asked about their ability to do certain ordinary tasks, such as taking care of themselves; ...

DETAILED DESCRIPTION:
The purpose of this study is to compare the clinical results of individuals living with advanced HIV infection who are treated with interleukin-2 (IL-2) plus active antiretroviral therapy (ART) to a control group of individuals treated with stable ART alone. The primary objective of the study is to determine if intermittent cycles of IL-2 delay the occurrence of opportunistic infections and the progression of advanced HIV disease compared to ART alone.

Patients will be assigned randomly to 1 of 2 groups. Patients in Group 1 will receive subcutaneous IL-2 twice a day for 5 days, every 8 weeks, in addition to ART. Patients in Group 2 will receive ART only. In both groups, CD4+ T cell counts and viral load are monitored.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects are eligible for this study if they have been on greater than or equal to 2 ART for greater than or equal to 4 months prior to randomization, with no change in the type of ART received during this 4-month period of time. For subjects who receive only 2 ART, at least one of these two medications should be a protease inhibitor (PI). Subjects are not eligible if ART is discontinued for a cumulative period of 7 or more days during the 4 months prior to randomization.

Subjects with documented HIV-1 infection. Acceptable documentation consists of either of the following:

Positive HIV-1 ELISA test and Western Blot;

Detectable plasma viral load measurement (greater than 500 RNA copies/mL using an ultrasensitive bDNA or PCR test or greater than 1500 RNA copies/mL using a non-ultrasensitive bDNA or PCR test).

CD4+ T cell counts: mean of 2 points obtained within 4 calendar months of randomization greater than or equal to 50 and less than 300 cells/mm(3). The first CD4+ count should be the most recent documented historical value and should be greater than or equal to 50 and less than 300 cells/mm(3); the second point should be pre-study visit 1.

Viral load less than 10,000 copies/mL, at 2 time points within 4 calendar months of randomization. The first viral load should be the most recent documented historical value and should be less than 10,000 copies/mL; the second time point should be pre-study visit 1.

Karnofsky performance status greater than or equal to 80%.

Age greater than or equal to 18 years old.

Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days prior to randomization. They must also understand that if they are randomized to the IL-2 group, they must practice effective contraception during their first 2 years of study participation. Pregnancy is discouraged among IL-2 recipients, but if an IL-2 recipient wishes to become pregnant after two years of trial participation she must alert the investigator prior to interruption of contraception. The potential for risk to the fetus must be carefully discussed with the subject before contraception is interrupted. Effective contraception will be continued for at least 24 hours following the interruption of IL-2 therapy. IL-2 will be held throughout the period of time during which the subject is not practicing effective birth control, throughout the pregnancy, and throughout any period of breast feeding. If oral contraceptive therapy is resumed after a period of interruption, IL-2 dosing will be delayed for 1 month following the reinstatement of oral contraceptive therapy. The subject must have a negative pregnancy test result prior to dosing with IL-2 after a lapse in effective contraception.

The following laboratory criteria must be fulfilled within 28 days of enrollment in the study:

Serum AST of less than or equal to 5 times upper limit of normal range (ULN);

Serum bilirubin less than or equal 2 times ULN (patients with Gilbert's syndrome or protease inhibitor-induced hyperbilirubinemia must have a serum bilirubin less than or equal to five times ULN);

Amylase less than 2.0 times ULN (hyperamylasemia that is determined to be non-pancreatic in origin does not necessarily constitute an exclusion to enrollment);

Less than 2 + proteinuria;

Serum creatinine less than or equal to 1.5 times ULN;

Absolute neutrophil count greater than or equal to 1000 cells/mm(3);

Hemoglobin of greater than or equal to 9.5 g/dL;

Platelet count of greater than or equal to 75,000/mm(3);

Negative HTLV-1 result.

Agree to participate in the study for 4.5 to 7.5 years.

Written informed consent.

EXCLUSION CRITERIA:

Certain AIDS-defining illnesses. These conditions include:

Patients with no prior history of AIDS-defining events are eligible for SILCAAT;

Patients with a prior medical history of one or more of the following AIDS-defining events are eligible only under the condition specified below:

Lymphoma (other than lymphoma of the brain): Patients with a history of successfully treated lymphoma are eligible, provided full remission was obtained at least 5 years prior to randomization. Full remission (or complete response) is defined as the absence of clinically detectable disease with normalization of any previously abnormal radiographic studies, and bone marrow examination. Patients with bone marrow positive lymphoma prior to chemotherapy must have had two repeat bone marrow examinations negative for lymphoma after chemotherapy at least 12 months prior to randomization.

Esophageal candidiasis; Patients with a prior history of successfully treated esophageal candidiasis are eligible if they have been free of clinical symptoms in the absence of antifungal suppressive therapy for at least 12 months prior to randomization. Documentation of a negative endoscopy should ideally be on record.

Invasive cervical cancer: Patients with a prior history of invasive cervical cancer are eligible if complete local cure of the cancer has been documented at least 5 years prior to randomization and there has been no evidence of metastatic disease at any time.

Kaposi's sarcoma: Patients are eligible if mucocutaneous lesions have been resolved or clinically stable for at least 12 months prior to randomization. Subjects with a history of visceral KS are excluded.

Mycobacterium tuberculosis or M. kansasii: Patients are eligible if clinical resolution of disease occurred at least 12 months prior to randomization and previously abnormal imaging studies have been normal, or stable after improvement, for at least 12 months prior to randomization. Documentation of microbiologic cure should ideally be on record. Therapy for tuberculosis or M. kansasii must have been completed at least 12 months prior to randomization.

Pneumocystis carinii pneumonia (PCP): Patients are eligible if clinical resolution of the disease occurred at least 12 months prior to randomization and previously abnormal imaging studies have been normal, or stable after improvement, for at least 12 months prior to randomization.

Recurrent pneumonia: Patients are eligible if there has been no evidence of pneumonia within 12 months prior to randomization.

Recurrent Salmonella septicemia: Patients are eligible if there has been no evidence of Salmonella septicemia within 12 months prior to randomization.

Wasting syndrome due to HIV: Patients are eligible for enrollment in SILCAAT if they have had a stable or increasing weight for at least 12 months prior to randomization.

Toxoplasmosis of the brain: Patients are eligible if their disease has been clinically resolved for at least 12 months prior to randomization. In addition, these patients must have a MRI or contrast CT scan of the brain performed within 1 month prior to randomization showing no sign of active disease.

Chronic intestinal cryptosporidiosis and chronic intestinal isosporiasis (greater than 1 month duration): Patients are eligible if their disease has been clinically resolved and they have been off specific therapy for at least 12 months prior to randomization. In addition, these patients must have at least one stool specimen documenting clearance of parasitic infection obtained within 1 month prior to randomization.

Patients with a history of any other AIDS-defining conditions as listed in the CDC 1993 Case Definition are not eligible for SILCAAT.

Subjects must not have clinically significant cardiac, pulmonary, thyroid, kidney or neurologic impairment, hemostasis disorder, or significant medical condition that would, in the opinion of the principal investigator, affect patient safety and/or compliance. In addition, subjects with the following conditions are specifically excluded: autoimmune disease, inflammatory bowel disease, psoriasis, optic neuritis, congestive heart failure, active ischemic heart disease, uncontrolled diabetes mellitus, moderate or severe hemophilia ( less than or equal to 5% of normal factor VIII levels), seizure disorder, uncontrolled hypothyroidism, cirrhosis and a prior medical history of transplantation. If an investigator has any reservations about the safety of enrolling a particular subject, he/she should consult with the medical monitor prior to screening the subject.

Psychiatric or cognitive disturbance or illness, or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect patient safety and/or compliance.

Malignancy requiring systemic chemotherapy within 12 months prior to randomization.

Current use or use within 4 weeks prior to randomization of systemic corticosteroid therapy or any agent, licensed or experimental, with known immunomodulatory effects (use of erythropoietin and anabolic steroids is allowed).

Current use, or use within 4 weeks of randomization of cytotoxic agents or antimetabolites; current use or use within 4 months of randomization of hydroxyurea or intravenous immunoglobulin.

Pregnant or lactating subjects.

Prior therapy with IL-2.

Prior participation in an ongoing IL-2 trial, eg, the ESPRIT trial.

Protocol non-compliance in a previous IL-2 trial.

Subjects with evidence of active acute infection within 2 weeks of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1695 (Actual)
Dates: Start 2001-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Neaton, PhD, Principal Investigator — University of Minnesota
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernstein ZP, Porter MM, Gould M, Lipman B, Bluman EM, Stewart CC, Hewitt RG, Fyfe G, Poiesz B, Caligiuri MA. Prolonged administration of low-dose interleukin-2 in human immunodeficiency virus-associated malignancy results in selective expansion of innate immune effectors without significant clinical toxicity. Blood. 1995 Nov 1;86(9):3287-94. PMID 7579429
- [Background] Autran B, Carcelain G, Li TS, Blanc C, Mathez D, Tubiana R, Katlama C, Debre P, Leibowitch J. Positive effects of combined antiretroviral therapy on CD4+ T cell homeostasis and function in advanced HIV disease. Science. 1997 Jul 4;277(5322):112-6. doi: 10.1126/science.277.5322.112. PMID 9204894
- [Background] Davey RT Jr, Chaitt DG, Piscitelli SC, Wells M, Kovacs JA, Walker RE, Falloon J, Polis MA, Metcalf JA, Masur H, Fyfe G, Lane HC. Subcutaneous administration of interleukin-2 in human immunodeficiency virus type 1-infected persons. J Infect Dis. 1997 Apr;175(4):781-9. doi: 10.1086/513971. PMID 9086130
- [Derived] Nordell AD, McKenna M, Borges AH, Duprez D, Neuhaus J, Neaton JD; INSIGHT SMART, ESPRIT Study Groups; SILCAAT Scientific Committee. Severity of cardiovascular disease outcomes among patients with HIV is related to markers of inflammation and coagulation. J Am Heart Assoc. 2014 May 28;3(3):e000844. doi: 10.1161/JAHA.114.000844. PMID 24870935
- [Derived] INSIGHT-ESPRIT Study Group; SILCAAT Scientific Committee; Abrams D, Levy Y, Losso MH, Babiker A, Collins G, Cooper DA, Darbyshire J, Emery S, Fox L, Gordin F, Lane HC, Lundgren JD, Mitsuyasu R, Neaton JD, Phillips A, Routy JP, Tambussi G, Wentworth D. Interleukin-2 therapy in patients with HIV infection. N Engl J Med. 2009 Oct 15;361(16):1548-59. doi: 10.1056/NEJMoa0903175. PMID 19828532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1971 participants were randomized at 139 sites in 11 countries. The first randomization was on 30 April 1999 and the last randomization was on 28 September 2002. Sites who re-consented 2/3 or more of their participants to Version 3 of the protocol were included in the analysis cohort. There are 1695 participants in the analysis cohort.
Groups:
- Proleukin Plus Antiretroviral Therapy: Patients receive an initial dose of 4.5 MIU of proleukin twice daily for 5 consecutive days every 8 weeks during the first year (6 cycles total). After the first year, additional cycles are given to either achieve or maintain the patient's CD4+ count goal. CD4+ goal is defined as an increase of 125 cells/cubic mm for participants in the 50-199 CD4+ count stratum, and an increase of 175 cells/cubic mm for participants in the 200-299 CD4+ stratum. In addition, all patients must be prescribed combination antiretroviral drug treatment. The choice of combination therapy is left to the discretion of the treating clinician. Investigators will use their national guidelines for determining when antiretroviral therapy should be changed and for when determining when therapy should be used. All patients must take antiretroviral therapy during each 5-consecutive-day treatment cycle.
- Antiretroviral Therapy Only: All patients must be prescribed combination antiretroviral drug treatment. The choice of combination therapy is left to the discretion of the treating clinician. Investigators will use their national guidelines for determining when antiretroviral therapy should be changed and for when determining when therapy should be used.
Period: Overall Study
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Started | 849 (138 were excluded from sites that did not re-consent 2/3 of patients to the amended protocol in 2003) | 846 (138 were excluded from sites that did not re-consent 2/3 of patients to the amended protocol in 2003)
Completed | 758 | 746
Not Completed | 91 | 100
Not completed — Lost to Follow-up | 91 | 100

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only | Total
Number analyzed (Participants) | 849 | 846 | 1695
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 841 | 838 | 1679
  >=65 years | 8 | 8 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 41.8 (8.7) | 42.0 (8.8) | 41.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 143 | 280
  Male | 712 | 703 | 1415
Region of Enrollment [Number; unit: participants]
  Belgium | 16 | 13 | 29
  Germany | 50 | 46 | 96
  Spain | 139 | 131 | 270
  France | 47 | 50 | 97
  Italy | 131 | 142 | 273
  Netherlands | 11 | 12 | 23
  Argentina | 85 | 85 | 170
  Australia | 62 | 64 | 126
  United States | 203 | 203 | 406
  Canada | 68 | 62 | 130
  Brazil | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: New or Recurrent Disease Progression Events, as Defined, or Death.
Description: Number of participants with fatal or non-fatal AIDS-related opportunistic disease or death from any cause.
  AIDS-related opportunistic disease includes CDC Category C 1993 definition plus the following diseases: Aspergillosis, invasive; Bartonellosis; Chagas disease of the CNS; Herpes zoster, multidermal; Leishmaniasis, visceral; Lymphoma, Hodgkin's; Microsporidiosis (> 1 month's duration); Nocardiosis; Penicillium marneffti, disseminated; Pneumocystis carinii, extrapulmonary; Rhodococcus equi disease.
Time Frame: From randomization to date last known to be alive or November 15, 2008, whichever is earlier
Measure: Number; unit: Participants
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Number analyzed (Participants) | 849 | 846
Participants | 110 | 119
Statistical Analysis 1: Comparison: Proleukin Plus Antiretroviral Therapy vs Antiretroviral Therapy Only; Null hypothesis was that event rates in two groups are equal. Study was designed with 80%, two-sided alpha=.05, assuming a 28% reduction in the hazard of opportunistic disease or death; Test type: Superiority or Other; p = 0.47, Regression, Cox; Stratification by CD4+ count stratum (50-199 or 200-299) and country of randomization; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.70 to 1.18]

2. Secondary Outcome: All-cause Mortality
Description: Number of participants who died.
Time Frame: From randomization to date last known to be alive or November 15, 2008, whichever is earlier
Measure: Number; unit: Participants
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Number analyzed (Participants) | 849 | 846
Participants | 81 | 77
Statistical Analysis 1: Comparison: Proleukin Plus Antiretroviral Therapy vs Antiretroviral Therapy Only; Test type: Superiority or Other; p = 0.73, Regression, Cox; Stratification by CD4+ stratum and country of randomization; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.77 to 1.44]

3. Secondary Outcome: New or Recurrent Disease Progression Events
Description: Number of participants with fatal or non-fatal AIDS-related opportunistic disease.
  AIDS-related opportunistic disease includes CDC Category C 1993 definition plus the following diseases: Aspergillosis, invasive; Bartonellosis; Chagas disease of the CNS; Herpes zoster, multidermal; Leishmaniasis, visceral; Lymphoma, Hodgkin's; Microsporidiosis (> 1 month's duration); Nocardiosis; Penicillium marneffti, disseminated; Pneumocystis carinii, extrapulmonary; Rhodococcus equi disease.
Time Frame: From randomization to date last known to be alive or November 15, 2008, whichever is earlier
Measure: Number; unit: Participants
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Number analyzed (Participants) | 849 | 846
Participants | 49 | 66
Statistical Analysis 1: Comparison: Proleukin Plus Antiretroviral Therapy vs Antiretroviral Therapy Only; Test type: Superiority or Other; p = 0.10, Regression, Cox; Stratification by CD4+ stratum and country of randomization; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.51 to 1.06]

4. Secondary Outcome: Grade 4 Clinical Events
Description: Grade 4 clinical events were defined as potentially life-threatening events (excluding opportunistic disease) requiring medical intervention.
Time Frame: From randomization to date last known to be alive or November 15, 2008, whichever is earlier
Population: The outcome is the number of participants experiencing at least one grade 4 event.
Measure: Number; unit: Participants
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Number analyzed (Participants) | 849 | 846
Participants | 203 | 186
Statistical Analysis 1: Comparison: Proleukin Plus Antiretroviral Therapy vs Antiretroviral Therapy Only; Test type: Superiority or Other; p = 0.35, Regression, Cox; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.90 to 1.34]

5. Secondary Outcome: CD4+ Cell Count
Description: Mean CD4+ cell count (cells per cubic mm) averaged over follow-up
Time Frame: Every 4 months from randomization through date last known to be alive or November 15, 2008, whichever was earliest .
Measure: Mean (Standard Error); unit: cells per cubic mm
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Number analyzed (Participants) | 849 | 846
cells per cubic mm | 345.1 (5.1) | 292.1 (4.1)
Statistical Analysis 1: Comparison: Proleukin Plus Antiretroviral Therapy vs Antiretroviral Therapy Only; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 53.0, 95% CI 2-sided [40.3 to 65.7], Standard Error of Mean 6.5

6. Secondary Outcome: New or Recurrent Serious Disease Progression Events or Death
Description: Number of participants with fatal or non-fatal serious AIDS-related opportunistic disease.
  A serious disease progression event is one of the following: progressive multifocal leukoencephalopathy (PML), lymphoma, Kaposi's sarcoma (visceral), AIDS dementia complex (ADC) stage II or higher, toxoplasmosis, histoplasmosis (systemic), cryptococcosis (systemic), disseminated Mycobacterium avium complex (MAC) disease, wasting syndrome, and cytomegalovirus (CMV) disease.
Time Frame: From randomization to date last known to be alive or November 15, 2008, whichever is earlier
Measure: Number; unit: Participants
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Number analyzed (Participants) | 849 | 846
Participants | 19 | 28

ADVERSE EVENTS:
Time Frame: From randomization to date last known to be alive or November 15, 2008, whichever is earlier
Description: Adverse events are defined as Grade 4 events not due to progression of HIV disease.
  Serious and/or other [non-serious) adverse events were not collected/assessed. Other Adverse Events were not collected.
Arm/Group | Proleukin Plus Antiretroviral Therapy | Antiretroviral Therapy Only
Serious Adverse Events (participants affected / at risk) | 203/849 | 186/846
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proleukin Plus Antiretroviral Therapy (N=849) | Antiretroviral Therapy Only (N=846)
Aneamias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 3 (5) | 6 (6)
Haemolyses and related conditions (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Platelet disorders (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Spleen, lymphatic and reticuloendothelial system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
White blood cell disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrythmias (Cardiac disorders) | 4 (5) | 4 (5)
Cardiac disorder signs and symptoms (Cardiac disorders) | 0 (0) | 1 (1)
Cornoary artery disorders (Cardiac disorders) | 20 (29) | 20 (24)
Heart failures (Cardiac disorders) | 3 (3) | 6 (13)
Myocardial disorders (Cardiac disorders) | 1 (1) | 2 (2)
Pericardial disorders (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac valve disorders (Cardiac disorders) | 2 (2) | 1 (2)
Renal and urinary tract disoerders congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Endocrine disorders of gonadal function (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid gland disorders (Endocrine disorders) | 0 (0) | 2 (3)
Ocular neuromuscular disorders (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernias and other adominal wall conditions (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diverticular disorders (Gastrointestinal disorders) | 1 (1) | 2 (2)
Exocrine pancreas conditions (Gastrointestinal disorders) | 6 (13) | 6 (7)
Gastrointestinal condictions NEC (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal haemorrhages NEC (Gastrointestinal disorders) | 13 (15) | 5 (10)
Gastrointestinal inflammatory conditions (Gastrointestinal disorders) | 4 (4) | 3 (5)
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 6 (8) | 5 (9)
Gastrointestinal stenosis and obstructions (Gastrointestinal disorders) | 5 (9) | 3 (3)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastrointestinal ulceration and perforation (Gastrointestinal disorders) | 5 (5) | 3 (3)
Gastrointestinal vascular conditions (Gastrointestinal disorders) | 7 (9) | 2 (3)
Peritoneal and retrooperationael conditions (Gastrointestinal disorders) | 2 (2) | 4 (4)
Body temperature conditions (General disorders) | 3 (4) | 2 (2)
General system disorders NEC (General disorders) | 6 (6) | 3 (4)
Fatal outcomes (General disorders) | 1 (1) | 0 (0)
Therapeutic and nontherapeutic effects (excl toxicity) (General disorders) | 1 (1) | 0 (0)
Bile duct disorders (Hepatobiliary disorders) | 0 (0) | 2 (3)
Gallbladder disorders (Hepatobiliary disorders) | 4 (4) | 7 (7)
Hepatic and hepatobiliary disorders (Hepatobiliary disorders) | 20 (26) | 10 (14)
Allergic conditions (Immune system disorders) | 1 (1) | 1 (1)
Immune disorders NEC (Immune system disorders) | 0 (0) | 1 (1)
Bacterial infectious disorders (Infections and infestations) | 14 (19) | 18 (20)
Fungal infectious disorders (Infections and infestations) | 1 (1) | 0 (0)
Infections - pathogen unspecified (Infections and infestations) | 28 (31) | 27 (30)
Mycobacterial infectious disorders (Infections and infestations) | 1 (1) | 0 (0)
Viral infectious disorders (Infections and infestations) | 11 (11) | 11 (16)
Bone and joint injuries (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Injuries NEC (Injury, poisoning and procedural complications) | 2 (3) | 5 (5)
Procedural and device related injuries and complications NEC (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Medications errors (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Chemical injury and poisoning (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gastrointestinal investigations (Investigations) | 1 (1) | 0 (0)
Hepatobiliary investigations (Investigations) | 0 (0) | 1 (1)
Lipid analyses (Investigations) | 0 (0) | 1 (1)
Metabolic, nutritional and blood gas investigations (Investigations) | 0 (0) | 1 (1)
Acid-base disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Appetite and general nutritional disorders (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Glucose metabolism disorders (incl diabetes mellitus) (Metabolism and nutrition disorders) | 4 (9) | 1 (1)
Purine and pyrimidine metabolism disorders (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bone disorders (excl congenital and fractuers) (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Joint disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (8)
Musculoskeletal and connective tissue deformities (incl intervertebral disc disorders) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Endocrine neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Gastrointestinal neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (9) | 10 (11)
Hepatic and biliary neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatobiliary neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Leukaemias (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Mesotheliomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Miscellaneuous and site unspecified neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Miscellaneous and site unspecified neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nervous system neoplasms malignant and unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal and urinary tract neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Reproductive neoplasms female malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Reproductive neoplasms male malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Respiratory and mediastinal neoplams malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (14) | 11 (13)
Skin neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (9) | 4 (5)
Oncologic complications and emergencies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system vascular disorders (Nervous system disorders) | 9 (9) | 8 (10)
Cranial nerve disorders (excl neoplasms) (Nervous system disorders) | 1 (1) | 3 (3)
Encephalopathies (Nervous system disorders) | 2 (2) | 2 (2)
Headaches (Nervous system disorders) | 2 (2) | 0 (0)
Movement disorders (incl parkinsonism) (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorders NEC (Nervous system disorders) | 0 (0) | 2 (2)
Neuromuscular disorders (Nervous system disorders) | 1 (1) | 0 (0)
Seizures (incl subtypes) (Nervous system disorders) | 3 (4) | 4 (4)
Spinal cord and nreve root disorders (Nervous system disorders) | 1 (1) | 1 (1)
Structural brain disorders (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety disorders and symptoms (Psychiatric disorders) | 3 (3) | 0 (0)
Cognitive and attention disorders and distrubances (Psychiatric disorders) | 1 (1) | 0 (0)
Deliria (incl confusion) (Psychiatric disorders) | 1 (1) | 1 (1)
Depressed mood disorders and disturbances (Psychiatric disorders) | 7 (8) | 4 (4)
Manic and bipolar mood disorders and disturbances (Psychiatric disorders) | 2 (2) | 0 (0)
Personality disorders and disturbances in behaviour (Psychiatric disorders) | 0 (0) | 1 (2)
Psychiatric disorders NEC (Psychiatric disorders) | 4 (5) | 0 (0)
Schizophrenia and other psychotic disorders (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal and self-injurious behaviours NEC (Psychiatric disorders) | 10 (11) | 4 (4)
Nephropathies (Renal and urinary disorders) | 1 (1) | 4 (4)
Renal disorders (excl nephropathies) (Renal and urinary disorders) | 5 (6) | 12 (13)
Urinary tract signs and symptoms (Renal and urinary disorders) | 2 (3) | 2 (2)
Urolithiases (Renal and urinary disorders) | 4 (6) | 3 (3)
Breast disorders (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervix disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Male reproductive tract infections and inflammations (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine, pelvic and broad ligament disorders (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Vulvovaginal disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchial disorders (excl neoplasms) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (6)
Thoracic disorders (excl lung and pleura) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract disorders (excl obstruction and infection) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pleural disorders (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pulmonary vascular disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (12)
Upper respiratory tract disorders (excl infections) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin and subcutaenous tissue disorders NEC (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Vascular therapeutic procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
Nervous system, skull and spine therapeutic procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
Hepatobiliary therapeutic procedures (Surgical and medical procedures) | 1 (1) | 1 (1)
Aneurysms and artery dissections (Vascular disorders) | 2 (3) | 0 (0)
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Vascular disorders) | 1 (1) | 2 (2)
Decreased and nonspecific blood pressure disorders and shock (Vascular disorders) | 3 (3) | 3 (4)
Embolism and thrombosis (Vascular disorders) | 4 (4) | 0 (0)
Vascular disorders NEC (Vascular disorders) | 1 (1) | 0 (0)
Vascular haemorrhagic disorders (Vascular disorders) | 1 (1) | 0 (0)
Vascular hypertensive disorders (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes